CLINICAL TRIAL: NCT02162680
Title: An Evaluation of the Effectiveness of Local Anesthetics Used During Intravenous Catheter Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00015861
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-06

CONDITIONS: IV Insertion Pain
Keywords: local anesthesia; intravenous catheter
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- lidocaine (Active Comparator): 1% lidocaine intradermal injection
  Interventions: Drug: 1% lidocaine
- bacteriostatic normal saline (BNS) (Active Comparator): bacteriostatic normal saline (BNS) injection
  Interventions: Drug: bacteriostatic normal saline (BNS)
- no local anesthetic (No Intervention): usual care practice of no local anesthetic administration

INTERVENTIONS:
Drug: 1% lidocaine
  Arms: lidocaine
Drug: bacteriostatic normal saline (BNS)
  Arms: bacteriostatic normal saline (BNS)

SUMMARY:
The purpose of this study is to compare how well different anesthetic, or numbing, solutions injected under the skin work in reducing the discomfort associated with placing a catheter in a vein. Two different medications, lidocaine and normal saline with benzyl alcohol, have been found to be effective in reducing discomfort when injected under the skin just prior to inserting the catheter. This study compares these two solutions, and will compare the discomfort that occurs both with and without using these solutions.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 or older)
* admitted to a general medical or surgical unit at Durham Regional Hospital (DRH)
* have a physician's order for an IV
* are able to speak, read and understand English
* referred to the Vascular Access Specialty Team (VAST) at DRH for IV catheterization

Exclusion Criteria:

* admission to the emergency room, pre-op unit, an outpatient unit, a psychiatric unit, an intensive care unit, a pre- or postnatal care unit, or labor and delivery units;
* history of a psychological disorder, as determined from the patient's chart;
* history of peripheral neuropathy, as determined by patient's chart;
* history of IV drug abuse, as determined from the patient's chart;
* decreased sensation in the arm or hands, as reported in the chart or by the patient;
* patient disorientation or confusion (i.e., unable to state person, place, time or unable to comprehend instructions for completing Visual Analog Scale);
* a known allergy to lidocaine or benzyl alcohol as determined from the patient's chart;
* veins that cannot be palpated and are difficult to visualize by VAST nurses;
* pregnancy;
* an order for the emergency insertion of an IV by the patient's doctor or assigned nurse;
* an IV insertion that requires the use of a catheter gauged 18 or larger
* severe vision impairment, as determined by the patient's inability to read the Visual Analogue Scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Aucoin, DNS, RN, Principal Investigator — Duke Health

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 99 subjects consented in the study. 1 subject withdrawn from study by PI, therefore 98 subjects completed study.
Groups:
- Lidocaine: 1% lidocaine intradermal injection
  1% lidocaine
- Bacteriostatic Normal Saline (BNS): bacteriostatic normal saline (BNS) injection
  bacteriostatic normal saline (BNS)
Period: Overall Study
Arm/Group | no Local Anesthetic | Lidocaine | Bacteriostatic Normal Saline (BNS)
Started | 33 | 33 | 32
Completed | 33 | 33 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | no Local Anesthetic | Lidocaine | Bacteriostatic Normal Saline (BNS) | Total
Number analyzed (Participants) | 33 | 33 | 32 | 98
Age, Customized [Number; unit: participants]
  18 and older | 33 | 33 | 32 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 23 | 16 | 55
  Male | 17 | 10 | 16 | 43
Race/Ethnicity, Customized [Number; unit: participants]
  White | 23 | 21 | 15 | 59
  African American | 8 | 7 | 15 | 30
  Other | 2 | 5 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 32 | 98

OUTCOME MEASURES:

1. Primary Outcome: Differences in Patients' Perceptions of Pain Between Treatment Methods
Description: The visual analog pain scale is a patient-reported measure of pain on a 10-point scale with 0 being no pain and 10 being worst possible pain. The visual analog pain score will be completed at the following time points: pre injection, during injection, and during catheter insertion.
Time Frame: at pre injection, during anesthetic injection, and during catheter insertion, up to approximately 1 minute
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | no Local Anesthetic | Lidocaine | Bacteriostatic Normal Saline (BNS)
Number analyzed (Participants) | 33 | 33 | 32
units on a scale
  Pain pre injection | 0.015 (0.87) | 0 (0) | 0 (0)
  Pain during catheter insertion | 1.909 (2.127) | 0.197 (0.499) | 0.609 (1.674)
  Pain during study drug injection | NA (NA) — Participants did not receive a study drug injection. | 0.727 (1.039) | 0.781 (1.263)

ADVERSE EVENTS:
Arm/Group | no Local Anesthetic | Lidocaine | Bacteriostatic Normal Saline (BNS)
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes